CLINICAL TRIAL: NCT06001736
Title: Seventh Cervical Nerve Transfer for Spastic Arm Paresis: a Prospective Analysis of Efficacy in Ischemic Vs. Hemorrhagic Stroke
Brief Title: Utility of CC7 Transfer in Stroke Subtypes
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Responsible Party: Principal Investigator, Jennifer Hong, Principal Investigator, Dartmouth-Hitchcock Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY02000583
Record Dates: First submitted 2023-08-14; First posted 2023-08-21 (Actual); Last update posted 2024-10-22 (Actual); Status verified 2024-10

CONDITIONS: Stroke, Ischemic; Stroke Hemorrhagic; Spastic Hemiparesis
MeSH Terms: conditions — Ischemic Stroke; Hemorrhagic Stroke; Hemiplegia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Contralateral C7 root transfer for the treatment of spastic hemiparesis. (Experimental): The C7 nerve root transfer will occur to the patients on this arm.
  Interventions: Procedure: Contralateral C7 root transfer for the treatment of spastic hemiparesis.

INTERVENTIONS:
Procedure: Contralateral C7 root transfer for the treatment of spastic hemiparesis. — Performing surgery to transfer the C7 nerve to treat stroke patients experiencing spastic hemiparesis.

SUMMARY:
The purpose of this study is to evaluate the limb functional improvement after contralateral C7 root transfer in stroke patients.

DETAILED DESCRIPTION:
Spastic limb paresis after stroke is a cause of long-term disability and reduction is quality of life, with loss of hand dexterity being especially prohibitive. In the recovery phase after initial injury, neural reorganization occurs and has been observed in both ipsilateral and contralateral hemispheres. Previous studies have identified contralesional (opposite to the side of the injury), in other words, ipsilateral, activation in the recovery of paretic hand function. However, this pathway of recovery is limited due to sparse connections between the ipsilateral hemisphere and the affected arm/hand. By establishing an anatomic connection between the ipsilateral hemisphere and the paretic arm with contralateral nerve transfer, compensatory capacity of the ipsilateral hemisphere is facilitated. This cross neck C7-C7 root transfer is an established procedure for the treatment of brachial plexus injuries and recently, for the treatment of spastic arm paresis in those with cerebral injury.

ELIGIBILITY:
Inclusion Criteria:

* History of ischemic or hemorrhagic stroke with resultant arm paresis that has ceased to improve within 1-5 years of rehabilitation.

Exclusion Criteria:

* pregnancy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 95 (Estimated)
Dates: Start 2022-03-13 (Actual); Primary Completion 2027-03-01 (Estimated); Study Completion 2027-03-01 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in arm function, as measured by the Fugl-Meyer upper-extremity scale. | 12 months with visits at baseline and months 2, 4, 8, and 12 months after surgery.
  The Fugl-Meyer is a widely used and highly recommended stroke-speciﬁc, performance-based measure of impairment with 5 domains and a possible 226 points.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Hong, Dr., Principal Investigator — Dartmouth-Hitchcock Medical Center
Locations (1):
- Dartmouth-Health, Lebanon, New Hampshire, United States